CLINICAL TRIAL: NCT07183215
Title: Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory Biomarkers in Osteoarthritis Genu
Acronym: ETCS
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Srinalesti Mahanani, Dr., National Institute of Health Research and Development, Ministry of Health Republic of Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 055/20/VI/EC/KEPK/STIKES RSBK
Record Dates: First submitted 2025-09-06; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
Keywords: Osteoathritis; Pain; TNF Alfa; Interleukin 1; C-Reactive Protein
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, we will conduct a 2-arm, double-blind (patient and investigational blinded) to assess efficacy, tolerability and safety curcuminoid versus placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Capsules containing curcuminoid from Tumeric Extract three times a day for 3 weeks
  Interventions: Drug: Curcuminoid Standardized Turmeric Capsules
- Control Group (Placebo Comparator): Capsules containing maltose three times a day for 3 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcuminoid Standardized Turmeric Capsules — Samples were made from extracted turmeric and then optimized. The capsule formulation is made from turmeric rhizome extract which contains 30 mg of curcuminoids per capsule. In the study, standardized curcuminoid turmeric extract was given in capsules at 30 mg 3 times a day for 3 weeks
  Arms: Intervention Group
Other: Placebo — The capsule formulation is made from maltose which contains 10 mg of curcuminoids per capsule. In the study, the capsule was given in capsules at 30 mg 3 times a day for 3 weeks.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if Curcuminoid Standardized Turmeric Capsules works to treat Osteoarthritis Genu in adults. It will also learn about the safety of Curcuminoid Standardized Turmeric Capsules. The main questions it aims to answer are:

* Does Curcuminoid Standardized Turmeric Capsules lower the pain, TNF-Alpha, Interleukin-1 and CRP in the blood?
* What medical problems do participants have when taking Curcuminoid Standardized Turmeric Capsules? Researchers will compare Curcuminoid Standardized Turmeric Capsules to a placebo to see if Curcuminoid Standardized Turmeric Capsules works to treat Osteoarthritis Genu.

Participants will:

* Take Curcuminoid Standardized Turmeric Capsules or a placebo every day for 3 weeks
* Visit the clinic once every week for checkups and tests
* Keep a diary of their symptoms and the number of times they use a rescue paracetamol

DETAILED DESCRIPTION:
Evaluate the efficacy, safety, and tolerability of standardized curcuminoid from turmeric extract to TNF-Alpha, Interleukin-1 and CRP in elderly patients with Osteoarthritis Genu. This research is also to evaluate the effect of acupressure and standardized curcuminoid from turmeric extract vs placebo at three weeks : Knee pain as measured by the VAS score. Study design is randomized controlled trial, double-blind to assess efficacy, tolerability, and safety curcuminoid versus placebo. Patients can be pre-screened for specific x-ray and laboratory parameters. Eligible subjects will enter the washout for one week following a screening visit. After the washout period, eligible subjects will be randomized and treated for three weeks. The total duration of the study is up to 5 weeks. The primary efficacy variable is the number of TNF-Alpha, Interleukin-1 and CRP in blood, collected at Week 4 to BL (i.e., change from BL in the number of Leukocytes at Week 4). It will be analyzed using the Wilcoxon signed-rank test or paired t-test and the Mann-Whitney U test or independent t-test. The significance level will be set at 0.05. All outcome measures will be recorded at baseline and after two weeks of intervention

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Osteoarthritis which confirmed by physical examination and x-rays
2. Experience pain with a Numeric Rating scale of 1-7
3. Must be able to swallow capsules
4. Must be able to carry out mobility without assistance or with minimal assistance

Exclusion Criteria:

1. Parkinson's disease
2. Dementia disease
3. Psychosis disease
4. Fractures
5. Joint dislocations
6. Cancer
7. Rheumatic diseases other than Osteoarthritis (rheumatoid arthritis)
8. Undergoing joint replacement therapy.
9. Analgesic dependent disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Secretion of TNF Alpha | 3 weeks
  TNF alpha is a cytokine, a protein that plays a role in the immune system and inflammation. TNF alpha is produced by various types of cells, particularly activated macrophages, and plays a role in various biological processes such as inflammation and immunity against infection.
  The cytokine TNF alpha is an essential mediator in increasing the inflammatory response, which can be detected in the blood plasma of patients with Osteoarthritis. The TNF alpha examination was conducted using the Enzyme Linked Immunosorbent Assay (ELISA) method on blood plasma
Secretion of the Interleukin-1 | 3 weeks
  Interleukin-1 is a pro-inflammatory cytokine that plays a key role in immune and inflammatory responses, produced primarily by macrophages. IL-1 can cause fever, increase blood vessel permeability, and trigger bone and cartilage damage.
  The cytokine Interleukin-1 is an essential mediator in increasing the inflammatory response, which can be detected in the blood plasma of patients with Osteoarthritis. The Interleukin-1 examination was conducted using the Enzyme Linked Immunosorbent Assay (ELISA) method on blood plasma
Secretion of C Reactive Protein | 3 weeks
  C-reactive protein (CRP) is a blood marker for inflammation in the body, produced by the liver in response to infection, injury, or autoimmune conditions. A simple blood test measures CRP levels, with higher concentrations indicating greater inflammation.
  C-reactive protein (CRP) is measured with a blood test to detect and monitor inflammation in your body. A blood sample is taken from a vein and analyzed in a laboratory to determine the CRP level. The results are reported in milligrams per liter (mg/L), and higher than normal levels indicate inflammation that may be caused by infection, injury, or a chronic condition.

SECONDARY OUTCOMES:
Change of Pain | 3 weeks
  Therapy effectiveness is the ability of a given treatment regimen to suppress several expected outcome indicators. Other outcome indicators were measured before starting therapy and after 3 weeks of therapy, including knee pain, as measured using a VAS score. Pain is expressed on a scale of 0 to 10, with higher numbers indicating more severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- GBI Ngadinegaran, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koroljevic ZD, Jordan K, Ivkovic J, Bender DV, Peric P. Curcuma as an anti-inflammatory component in treating osteoarthritis. Rheumatol Int. 2023 Apr;43(4):589-616. doi: 10.1007/s00296-022-05244-8. Epub 2022 Nov 17. PMID 36394597
- [Background] Mahanani S, Kertia N, Madyaningrum E. Combination of Curcuminoids and Acupressure for Inflammation and Pain in Older People with Osteoarthritis Genu: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 24;13:e54970. doi: 10.2196/54970. PMID 38771152

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT07183215/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT07183215/ICF_001.pdf